CLINICAL TRIAL: NCT02914041
Title: Kyphotic Measure Using Distance From the Wall: Reliability, Validity and Distance From the Wall to Indicate Risk for Spinal Fracture
Brief Title: Kyphotic Measure Using Distance From the Wall
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Other Study IDs: PHD57I0037
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-09

CONDITIONS: Kyphosis
Keywords: Kyphosis; Kyphosis wall distance; elderly
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kyphosis group: Subjects are community-dwelling elderly with different degrees of kyphosis, aged at least 60 years with a body mass index between 18.5-29.9 kg/m2 and OWD >0 cm.

SUMMARY:
Are the KypDisT and conventional C7WD are practical, valid, reliable, and effectiveness of the tools to discriminate the functional ability impairments relating to kyphosis when compare with gold standard (Cobb's method), and compare among physical therapy, VHS and caregiver?

DETAILED DESCRIPTION:
1. To further develop an innovation to measure kyphosis using distance from the wall, a Kyphosis wall distance tool (KypDisT).
2. investigate validity of the measurements in terms of 2.1 Concurrent validity of conventional C7WD and KypDisT as compared to a gold standard (Cobb's method).

   2.2 Discriminative ability of conventional C7WD and KypDisT on functional abilities in elderly with different severity of kyphosis.
3. To investigate the reliability of the measurements in terms of 3.1 Test-retest reliability of conventional C7WD and KypDisT. 3.2 Reliability of conventional C7WD and KypDisT comparing among physical therapy, VHS and caregiver.
4. To explore the distance to indicate risk of spinal fracture to indicate a risk of spinal fracture.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling elderly with different degrees of kyphosis,
* Aged at least 60 years
* Body mass index between 18.5-29.9 kg/m2
* OWD >0 cm.

Exclusion Criteria:

* Present signs and symptoms that may affect participation in the study, i.e. unstable medical condition, pain or inflammation in the joints of the lower extremity (pain scale > 5), having sequelae of neurological deficits
* Unable to understand and follow a simple command used in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly who live community-dwelling with different degrees of kyphosis, aged at least 60 years with a body mass index between 18.5-29.9 kg/m2 and OWD >0 cm. (Wongsa et al., 2012). However, elderly are excluded if they present signs and symptoms that may affect participation in the study, i.e. unstable medical condition, pain or inflammation in the joints of the lower extremity (pain scale > 5), having sequelae of neurological deficits, and unable to understand and follow a simple command used in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
KMD | 7 days
  Kyphosis assessments using distance from the wall

SECONDARY OUTCOMES:
10MWT | 1 day
  walking speed
FTSST | 1 day
  Lower limb muscle strength
TUGT | 1 day
  Balance control
6MinWT | 1 day
  Walking endurance

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, PhD, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No